CLINICAL TRIAL: NCT03455673
Title: Diagnostic Accuracy of the ATE Score for the Exclusion of Intra-atrial Thrombi Before Catheter Ablation of Atrial Fibrillation: a Confirmatory Study
Brief Title: Exclusion of Intra-atrial Thrombus Before Catheter Ablation
Acronym: EXTRALUCID
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: Diagnostica Stago (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017/P02/211
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; Thrombi
MeSH Terms: conditions — Atrial Fibrillation; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral blood sample is collected for d-dimer assay at the inclusion. Frozen samples will be used to constitute a plasma bank to further confirm the study performances with other D-dimer assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial fibrillation: ATE score will be determined for patients hospitalized for ablation of atrial fibrillation or symptomatic left atrial tachycardia
  Interventions: Diagnostic Test: ATE score

INTERVENTIONS:
Diagnostic Test: ATE score — The Atrial Thrombus Exclusion (ATE) combine thromboembolic risk factors (hypertension, cardiac insufficiency, history of stoke) and d-dimer level for the prediction of intra-atrial thrombus :
  Hypertension = 1 Heart failure = 1 History of stroke = 1 High plasma d-dimer level (> 270 ng/ml) = 1

SUMMARY:
Atrial fibrillation is the most frequent heart rhythm disorder. Its symptomatic forms, resistant to drug therapy, require invasive management (catheter ablation), which exposes to potentially serious complications including thromboembolic complications. Despite anticoagulant treatment, intra-atrial thrombus, which is a contraindication to catheter ablation, is detected in nearly 2 % of cases. Its diagnosis requires prior transoesophageal echocardiography, an unpleasant examination.

A previous study (NCT02199080) showed that a zero ATE score, defined by no heart failure, no hypertension, no history of stroke, d-dimer < 270 ng/mL, has a negative predictive value of 100 % for the exclusion of intra-atrial thrombus.

The objective of the study is to confirm the negative predictive value, sensitivity and specificity of the ATE score for the exclusion of intra-atrial thrombus.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,
* Patients hospitalized for ablation of atrial fibrillation or symptomatic left atrial tachycardia,
* have signed or orally given an informed consent

Exclusion Criteria:

* Contraindication to transoesophageal echocardiography,
* Transoesophageal echocardiography made in another centre than the centre of ablation,
* Pregnant women, parturient mothers and nursing mothers,
* Lives in an institution on court or authority order,
* Severely altered psychological health,
* Persons leaving in health or social establishment,
* Minors,
* Under guardianship,
* Persons unable to give their consent,
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each centre, patient eligible for atrial fibrillation or left flutter ablation will be screened. In agreement with the physician performing the procedure, the study will be explained and proposed to the eligible patients by an investigator at the admission or at the pre-ablation consultation. It is strongly recommended to include patients consecutively in order to limit selection bias.
Sampling Method: Non-Probability Sample
Enrollment: 3160 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine MILHEM, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (15):
- France (14):
  - Service de cardiologie, Centre Hospitalier du pays d'Aix, Aix-en-Provence
  - Service de cardiologie, CH Annecy Genevois, Annecy
  - Service de cardiologie, CHU Brest, Brest
  - Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle
  - Service de cardiologie, CH Le Mans, Le Mans
  - Service de cardiologie, CHR Metz Thionville, Metz
  - Service de cardiologie, Hôpital privé du Confluent, Nantes
  - Service de cardiologie, CHU Nîmes, Nîmes
  - Hôpital Pitié Salpêtrière, Paris
  - Centre Hospitalier de Pau, Pau
  - Service de cardiologie, CHU Rouen, Rouen
  - Service de cardiologie, CHU Saint Etienne, Saint-Etienne
  - Service de cardiologie, CHU Toulouse, Toulouse
  - Service de cardiologie, Clinique Saint Joseph, Trélaze
- University Hospital Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Milhem A, Ingrand P, Treguer F, Cesari O, Da Costa A, Pavin D, Rivat P, Badenco N, Abbey S, Zannad N, Winum PF, Mansourati J, Maury P, Bader H, Savoure A, Sacher F, Andronache M, Allix-Beguec C, De Chillou C, Anselme F; ATE Study Group. Exclusion of Intra-Atrial Thrombus Diagnosis Using D-Dimer Assay Before Catheter Ablation of Atrial Fibrillation. JACC Clin Electrophysiol. 2019 Feb;5(2):223-230. doi: 10.1016/j.jacep.2018.09.009. Epub 2018 Nov 1. PMID 30784695
- [Background] Gage BF, Waterman AD, Shannon W, Boechler M, Rich MW, Radford MJ. Validation of clinical classification schemes for predicting stroke: results from the National Registry of Atrial Fibrillation. JAMA. 2001 Jun 13;285(22):2864-70. doi: 10.1001/jama.285.22.2864. PMID 11401607
- [Background] Natale A, Mohanty S, Goldstein L, Gomez T, Hunter TD. Real-world safety of catheter ablation for atrial fibrillation with contact force or cryoballoon ablation. J Interv Card Electrophysiol. 2021 Apr;60(3):445-452. doi: 10.1007/s10840-020-00734-w. Epub 2020 May 11. PMID 32390061
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Scherr D, Dalal D, Chilukuri K, Dong J, Spragg D, Henrikson CA, Nazarian S, Cheng A, Berger RD, Abraham TP, Calkins H, Marine JE. Incidence and predictors of left atrial thrombus prior to catheter ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2009 Apr;20(4):379-84. doi: 10.1111/j.1540-8167.2008.01336.x. Epub 2008 Oct 27. PMID 19017348
- [Background] Puwanant S, Varr BC, Shrestha K, Hussain SK, Tang WH, Gabriel RS, Wazni OM, Bhargava M, Saliba WI, Thomas JD, Lindsay BD, Klein AL. Role of the CHADS2 score in the evaluation of thromboembolic risk in patients with atrial fibrillation undergoing transesophageal echocardiography before pulmonary vein isolation. J Am Coll Cardiol. 2009 Nov 24;54(22):2032-9. doi: 10.1016/j.jacc.2009.07.037. PMID 19926009

RESULTS

PARTICIPANT FLOW:
Groups:
- Atrial Fibrillation: ATE score will be determined for patients hospitalized for ablation of atrial fibrillation or symptomatic left atrial tachycardia
  ATE score: The Atrial Thrombus Exclusion (ATE) combine thromboembolic risk factors (hypertension, cardiac insufficiency, history of stoke) and d-dimer level for the prediction of intra-atrial thrombus :
  Hypertension = 1 Heart failure = 1 History of stroke = 1 High plasma d-dimer level (> 270 ng/ml) = 1
Period: Overall Study
Arm/Group | Atrial Fibrillation
Started (Potentially eligible patients) | 3160
Patients With an ATE Score | 3099
Completed | 3072
Not Completed | 88

BASELINE CHARACTERISTICS:
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 3072
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1422
  >=65 years | 1650
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 863
  Male | 2209
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 2996
  Switzerland | 76
Clinical history of heart failure [Count of Participants; unit: Participants] | 459
Clinical history of stroke or transient ischemic attack [Count of Participants; unit: Participants] | 175
Hypertension [Count of Participants; unit: Participants] | 1292
Diabetes mellitus [Count of Participants; unit: Participants] | 350
Vascular disease [Count of Participants; unit: Participants] | 376
CHA2DS2VASc score [Median (Inter-Quartile Range); unit: units on a scale] — CHA2DS2VASc score is a stroke risk stratification scheme based on a risk factor approach
  Risk factors are quoted as follow:
  * Congestive heart failure and/or left ventricular ejection fraction ≤ 40% =1
  * Hypertension=1
  * Age ≥ 75=2
  * Diabetes mellitus=1
  * Stroke and/or transient ischemic attack and/or thromboembolism=2
  * Vascular disease=1
  * Age 65-74=1
  * Female=1
  Score range from 0 (lowest risk factor) to 10 (highest risk factor)
  units on a scale | 2 [1 to 3]
CHADS2 score [Median (Inter-Quartile Range); unit: units on a scale] — CHADS2 score is a stroke risk stratification scheme based on a risk factor approach
  Risk factors are quoted as follow:
  * Congestive heart failure=1,
  * Hypertension=1,
  * Age > 75=1
  * Diabetes mellitus=1,
  * Stroke or transient ischemic attack=1
  Score range from 0 (lowest risk factor) to 5 (highest risk factor)
  units on a scale | 1 [0 to 1]
Diagnosis [Count of Participants; unit: Participants]
  Left atrial tachycardia | 308
  Paroxysmal fibrillation | 1638
  Persistent fibrillation | 1126

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Atrial Thrombus and a Zero ATE Score
Description: Patients with atrial thrombus diagnosed by pre-procedural transoesophageal echocardiography, without hypertension, heart failure, history of stroke and a plasma d-dimer level < 270 ng/ml ATE : Atrial Thrombus Exclusion minimum value = 0 maximum value = 4, patient at higher risk of atrial thrombus
Time Frame: at most 48 hours before ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 3072
Participants
  ATE = 0, thrombus | 2
  ATE = 0, No thrombus | 816
  ATE > 0, thrombus | 27
  ATE > 0, No thrombus | 2227

2. Secondary Outcome: Number of Patients With Atrial Thrombus
Description: Patients with atrial thrombus diagnosed by pre-procedural transoesophageal
Time Frame: at most 48 hours before ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 3072
Participants
  Thrombus diagnosed by the reference method | 29
  No thrombus diagnosed by the reference method | 3043

3. Secondary Outcome: Number of Patients With Atrial Thrombus Among Patients With a Zero CHADS2VASC Score
Description: Patients with atrial thrombus diagnosed by pre-procedural transoesophageal echocardiography, and without congestive heart failure, hypertension, diabetes mellitus, vascular disease [previous myocardial infarction, peripheral arterial disease or aortic plaque], history of stroke or transient ischemic attack, aged under 75, and male minimum value = 0 maximum value = 10, at most risk of stroke
Time Frame: at most 48 hours before ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 3072
Participants
  CHADS2VASC = 0, thrombus | 3
  CHADS2VASC = 0, no thrombus | 604
  CHADS2VASC > 0, thrombus | 26
  CHADS2VASC > 0, no thrombus | 2438
  CHADS2VASC score unavailable | 1

4. Secondary Outcome: Number of Patients With Atrial Thrombus Among Patients With a Zero CHADS2 Score
Description: Patients with atrial thrombus diagnosed by pre-procedural transoesophageal echocardiography, and without congestive heart failure, hypertension, diabetes mellitus, history of stroke or transient ischemic attack, and aged under 75 minimum value = 0 maximum value = 6, at most risk of stroke
Time Frame: at most 48 hours before ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 3072
Participants
  CHADS2 = 0, thrombus | 4
  CHADS2 = 0, no thrombus | 1285
  CHADS2 > 0, thrombus | 25
  CHADS2 > 0, no thrombus | 1757
  CHADS2 score unavailable | 1

ADVERSE EVENTS:
Time Frame: The study lasted 48 hours for each participant. Adverse events were collected during these 48 hours.
Arm/Group | Atrial Fibrillation
All-Cause Mortality (participants affected / at risk) | 0/3072
Serious Adverse Events (participants affected / at risk) | 2/3072
Other Adverse Events (participants affected / at risk) | 1/3072
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atrial Fibrillation (N=3072)
Pericarditis (Cardiac disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atrial Fibrillation (N=3072)
Loss of consciousness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT03455673/Prot_SAP_000.pdf